CLINICAL TRIAL: NCT04147624
Title: REACTION Trial: Medical Nutrition in Cognitive Aging, a Double-blind Controlled 6-month Study
Brief Title: Reducing the Effects of Aging on Cognition With Therapeutic Intervention of an Oral Nutrient (REACTION): A Pilot Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: American Academy of Neurology (Other)
Responsible Party: Principal Investigator, Christian Camargo, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20190750
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Decline
Keywords: Memory; Cognitive Aging
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Souvenaid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Participants in the treatment group will receive 125 mL of Souvenaid taken by mouth, once daily, for 6 consecutive months.
  Interventions: Drug: Souvenaid
- Placebo Group (Placebo Comparator): Participants in the treatment group will receive 125 mL of iso-caloric placebo taken by mouth, once daily, for 6 consecutive months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Souvenaid — Souvenaid is an oral beverage that contains a vitamin mixture (Vitamin A, B1, B2, B3, B5, D) plus three main active ingredients: omega-3 fatty acids, uridine monophosphate, and choline.
  Arms: Treatment Group
Other: Placebo — The Placebo used in this study is an oral beverage vitamin mixture containing Vitamins A, B1, B2, B3 and B5.
  Arms: Placebo Group

SUMMARY:
The purpose of this research is to assess the feasibility (e.g., recruitment rate, adherence rate and retention rate) of a clinical trial using virtual assessments to investigate the effect of a 6-month administration of a specific multi-nutrient oral supplement on cognitive aging.

The study will also test whether a 6-month daily intake of a specific multinutrient can delay or reverse the effects of normal cognitive aging on other cognition domains as well as quality of life as measured by virtual assessments.

DETAILED DESCRIPTION:
Participants with cognitive aging who meet the eligibility criteria are provided study information and scheduled for a screening visit via virtual encounter. At the screening visit, participants meeting criteria are enrolled, and a baseline visit is scheduled (same day, or separately.) The participants are then randomized to either the test product (specific multi-nutrient) or placebo. Study parameters will be assessed at baseline, and 6 months via a virtual online platform. Patients will be contacted monthly via telephone to promote compliance and monitor progress. An optional sample of blood may be provided by the participant if willing to participated in this optional sub-study.

ELIGIBILITY:
Inclusion Criteria:

1. English or Spanish speaking participants considered to have age-related cognitive decline based on the following criteria:

   A) RBANS (Verbal Memory Retention) A score ≥70% on list learning retention AND ≥80% on story memory retention and B) Subjective Cognitive Decline (SCD) 9-item brief screening tool score within the 25th percentile (SCD =1) and 75th percentile (SCD = 6) and C) MoCA ≥24
2. Age 55-89
3. Written informed consent provided by participant

Exclusion Criteria:

1. Enrollment in any other clinical trial within 30 days prior to participation
2. Major Neurocognitive Disorder ("Dementia") according to the Diagnostic and Statistical Manual of Mental Disorders 5th Edition and/or NIAA Criteria
3. Use of any AD medication (e.g., cholinesterase inhibitors, NMDA antagonists), or OTC supplements or cognitive/memory enhancers
4. Use of omega-3 fatty acids in the 30 days prior to participation
5. Intake of Vitamins B6 and B12, folate, Vitamins C and E > 300% RDI in the 24 days prior to participation
6. Concurrent major medical or neurological illness
7. Prior clinical history of stroke
8. History of substance abuse (e.g., alcohol, drugs)
9. Untreated Major Depressive Disorder that has not been in remission for at least 6 months prior to participation

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Successful recruitment rate | Baseline
  50% or more of those who fulfill the criteria and are invited to participate
Successful recruitment time | Baseline
  <110% of planned time
Successful adherence to the intervention | 6 months
  80% or more of the test product is consumed
Successful Retention rate | 6 months
  Less than 30% of the participants drop-out; Tracking the percentage of participants in the "Per-Protocol" population (i.e., no protocol deviation) less than 30% of the participants drop-out
  Tracking the percentage of participants in the "Per-Protocol" population (i.e., no protocol deviation)
Overall feasibility of this study will be assessed | 6 months
  Will take into account all feasibility parameters

SECONDARY OUTCOMES:
Rey Auditory Verbal Learning Task (RAVLT) or WHO/UCLA Auditory Verbal Learning Task (AVLT) | Baseline, 6 months
  The test takes 10-15 minutes plus a 30-minute delay during which time other measures can be done.
Digit Span (WAIS-IV) | Baseline, 6 months
  measures attention and working memory using exercises that require participants to recite a A series of progressively longer sequence of numbers in forwards, backwards and sequencing order.
The Oral Trail Making Test B | Baseline, 6 months
  (TMT-B) assesses working memory and cognitive flexibility. Participants are asked to verbally alternate between letters and numbers in sequential order as quickly as possible.
Matrix reasoning from the Test My Brain (TMB) research battery | Baseline, 6 months
  The task provides a measure of fluid intelligence and non-verbal reasoning. It is based on a well-validated and widely used matrix reasoning tasks but adapted for virtual administration.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Camargo, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No